CLINICAL TRIAL: NCT01978535
Title: A Randomized, Controlled, Double Blinded Clinical Trial of Intravenous Iron Sucrose in Adolescents With Non-anemic Iron Deficiency and Postural Orthostatic Tachycardia Syndrome (POTS)
Brief Title: Iron Sucrose in Adolescents With Iron Deficiency and Postural Orthostatic Tachycardia Syndrome (POTS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruiting subjects.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amie E. Jones, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-009963
Record Dates: First submitted 2013-06-07; First posted 2013-11-07 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Ferric Oxide, Saccharated; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron infusion (Experimental): Iron Sucrose (Venofer (R))
  Interventions: Drug: Iron infusion
- Normal saline infusion (Placebo Comparator): Equal volume to intervention of normal saline
  Interventions: Drug: Normal saline infusion

INTERVENTIONS:
Drug: Iron infusion — 5 mg/kg of intravenous iron sucrose supplied as Venofer (TM) with a maximum dose of 200mg. Iron sucrose will be diluted to 1 mg of elemental iron in 1 mL of NaCl 0.9% with a maximum volume of 210 mL.
  Other Names: Iron sucrose; Venofer (TM)
  Arms: Iron infusion
Drug: Normal saline infusion — Normal saline (NaCl 0.9%) 5 mL/kg up to a maximum volume 210 mL
  Other Names: Normal saline; NaCl 0.9%
  Arms: Normal saline infusion

SUMMARY:
This study is designed to investigate whether the treatment of non-anemic iron deficiency with intervenous iron sucrose will result in decreased symptom reporting and improved cardiovascular indices in adolescents (age 12-21) with Postural Orthostatic Tachycardia Syndrome (POTS).

DETAILED DESCRIPTION:
Postural orthostatic tachycardia syndrome (POTS) is characterized by an exaggerated heart rate response to the standing position in a patient with symptoms of orthostatic intolerance. It is likely a heterogeneous disorder representing a common manifestation of a number of possible underlying derangements such as impaired sympathetically mediated vasoconstriction, excessive sympathetic drive, volume dysregulation and deconditioning. While the actual prevalence of POTS is unknown, it has been estimated to affect at least 500,000 individuals in the United States. It predominately affects young individuals, and particularly women.

The prevalence of iron deficiency in adolescents with POTS has been reported to be greater than that expected in the general adolescent population. The use of intravenous iron sucrose has been shown to be a safe and effective therapy for correcting iron deficiency in children and adolescents. Anecdotal experience at our clinic has demonstrated an immediate reduction in self-reported orthostatic symptoms in several patients diagnosed with POTS following the administration of intravenous iron sucrose for iron deficiency.

This study is a randomized, double blind, placebo-controlled study to assess the efficacy of a single iron sucrose infusion in adolescents with non-anemic iron deficiency and POTS. Subjects will be screened at outpatient clinic visit appointments. Interested qualified subjects will be consented and offered participation in this trial. Once consent and assent (for patients less than 18 years of age) has been obtained, subjects will be randomized to either treatment or placebo group. Subjects will participate in two on site study visits. During the first visit subjects will complete baseline laboratory studies, tilt table test and study questionnaires. Subjects will then receive the intervention study drug or placebo. The second study visit will occur 7 days + 2 days from the first study visit. During the second study visit subjects will repeat laboratory studies, tilt table test and study questionnaires. Follow up questionnaires will be sent to all subjects six months following the initial study visit.

ELIGIBILITY:
Inclusion criteria

* aged 12-21 years
* chronic (>3 months)symptoms of orthostatic intolerance (including but not limited to lightheadedness, syncope, headache, fatigue, weakness, sweating, nausea and palpitations)
* symptomatic orthostatic heart rate increase of greater than or equal to 40 beats per minute during a 10 minute 70 degree head up tilt study
* presence of non-anemic iron deficiency, defined as serum ferritin level less than or equal to 20 ug/L with normal hemoglobin

Exclusion criteria

* orthostatic hypotension within 3 minutes of 70 degree head up tilt
* pregnant or lactating females
* presence of other organ failure or systemic illness that can affect autonomic function
* concurrent medication therapy with anticholinergic, alpha-adrenergic antagonists, beta-adrenergic antagonists unless medication is held for five half-lives prior to study
* laboratory evidence of anemia or iron overload
* personal history of hematochromatosis or first degree relative with hematochromatosis
* known sensitivity to Venofer (TM) or other intravenous iron preparations

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amie Jones, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic, Rochester, Minnesota.
Period: Overall Study
Arm/Group | Iron Infusion | Normal Saline Infusion
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Infusion | Normal Saline Infusion | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Indices-interval Change in Heart Rate During 10-minute Head up Tilt Table Test
Description: This study will assess whether a single infusion of iron sucrose will improve cardiovascular indices, specifically a reduction in the interval of measured heart rate change, during a ten minute head up tilt, in adolescent subjects with POTS and non-anemic iron deficiency
Time Frame: 7 (+/- 2) days following intervention
Population: The outcome measure was not analyzed because there were insufficient data.
Arm/Group | Iron Infusion | Normal Saline Infusion
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Six months
Arm/Group | Iron Infusion | Normal Saline Infusion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulty in recruiting subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT01978535/Prot_SAP_000.pdf